CLINICAL TRIAL: NCT07041905
Title: Effects of Total and Selective Caries Removal - Requiring or Avoiding Vital Pulp Therapy - on Pulp Vitality and Postoperative Pain in Deep Carious Mature Permanent Teeth: A Split-Mouth Clinical Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Zehra SUSGUN YILDIRIM, Principal Investigator, Cukurova University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: D-SCR-2025-01
Record Dates: First submitted 2025-06-19; First posted 2025-06-27 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-06

CONDITIONS: Pulp Exposure, Dental; Deep Dental Caries
MeSH Terms: conditions — Dental Pulp Exposure

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients and outcome assessors were blinded to the intervention groups. The operator was not blinded due to the visible differences between total and selective caries removal techniques.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (Active Comparator): Complete caries excavation
  Interventions: Procedure: Total Caries Removal
- Arm 2 (Experimental): Partial caries excavation
  Interventions: Procedure: Selective Caries Removal

INTERVENTIONS:
Procedure: Total Caries Removal — Arm 1: "Total caries removal (complete excavation to hard dentin)"
  Arms: Arm 1
Procedure: Selective Caries Removal — Partial removal leaving affected dentin near pulp.
  Arms: Arm 2

SUMMARY:
The effect of selective caries cleaning and total caries cleaning on pulp health and post operative pain in teeth with deep caries will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥15 years with bilateral deep carious mature permanent teeth.
* Positive vitality test (cold sensitivity).
* No spontaneous pain or periapical radiolucency.
* Willingness to attend 6- and 12-month follow-ups

Exclusion Criteria:

* Uncontrolled systemic diseases Pregnancy or allergy to dental materials used Teeth with irreversible pulpitis (spontaneous pain, necrosis) Non-restorable teeth (fractures, extensive decay)

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Early postoperative pain intensity (VAS) after total vs. selective excavation | first week
  The patient will be asked to rate his/her pain on day 1, 3 and 7 according to VAS
dentin bridge formation | twelve months
  no dentin bridge formation is expected in selective caries cleaning, while dentin bridge formation will be observed radiologically in total cleaning
pulp survival at twelve months | twelve months
  The pulp is expected to remain vital, with no percussion tenderness and no spontaneous pain

CONTACTS AND LOCATIONS:
Locations (1):
- Cukurova University, Adana, Turkey (Türkiye)